CLINICAL TRIAL: NCT05531396
Title: The Effects of Agility Training and Its Relations on Physical Performance, Cognitive Function and Brain Activities in Elderly
Brief Title: Agility Training on Physical Performance, Cognitive Function and Brain Activities in Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202205012RINC
Record Dates: First submitted 2022-08-05; First posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-05

CONDITIONS: Elderly; Healthy
Keywords: Agility training; Physical function; Cognition function; Elderly; Functional near-infrared spectroscopy (fNIRS)

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Education (Active Comparator)
  Interventions: Other: Health Education
- Agility Training Group (Experimental)
  Interventions: Other: Agility Training

INTERVENTIONS:
Other: Agility Training — Participants will receive 60 minutes of exercise, twice a week, for a total of 8 weeks, and training will be conducted by a well-trained physical therapist. The intervention will comprise a 5-minute warm-up, 45 minutes of main exercise, and a 10-minute cool-down period, for a total of 60 minutes each session. During the warm-up and cool-down, participants will do static and dynamic whole-body stretching exercises.
  Arms: Agility Training Group
Other: Health Education — Participants in the control group will receive health educational guidelines. Guideline contents include home-based exercise program, nutrition recommendations, and fall prevention education. The home-based exercise program will emphasize how to safely and properly perform stretching and whole-body exercises.
  Arms: Health Education

SUMMARY:
Agility comprised of cognitive and physical functions, which influences whole-body movement with change of speed and direction. Agility training is widely used in athletes, and recent studies have begun to apply it into the elderly. Agility training is multidimensional and highly functional, which makes it possible to provide more efficient training in limited time. In elderly, the decrement of cognitive function, muscle strength in the upper and lower limbs, the percentage of body fat, body flexibility and endurance caused by aging will make it difficult for the elderly to perform movements. Therefore, it is essential to explore whether agility training can achieve the improvement of the physical function and cognitive function in elderly, and to find the relationship between the two functions and brain activity. Method: This study will recruit 60 participants, and randomly allocate to control group and agility training. The training groups will have 8 weeks of training, 2 times a week, 45 minutes of training each time. Assessment will be performed before and after intervention in 1-week, and with 1-month follow-up. Assessment including agility ability, physical function, cognitive function, brain activity, and functional assessment scales.

ELIGIBILITY:
Inclusion Criteria:

1. older than 65 years old
2. score of Mini-Mental State Examination (MMSE) ≥ 24
3. able to walk independently for more than 30 meters without assistive aids
4. able to follow orders

Exclusion Criteria:

1. poorly controlled or unstable systematic disease
2. has a history of central nervous system disease
3. currently taking antidepressants, anti-anxiety, or other psychiatric drugs that may affect blood flow in the brain
4. has other medical conditions for which exercise is contraindicated; (5) subjects with achromatopsia.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-05 (Estimated); Primary Completion 2023-05-23 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Agility Challenge for the Elderly (ACE) | Baseline, 8 weeks, and 12 weeks
  An agility course developed for a 9m x 18m volleyball court and includes three segments that each aim to test a specific aspect of agility, including stop-and-go, change of direction, and spatial orientation.

SECONDARY OUTCOMES:
Fall history and fear of falls | Baseline, 8 weeks, and 12 weeks
  Fall history will be recorded by the number of fall episodes in the past 6 months and whether it caused injury.
Quality of life (QOL) | Baseline, 8 weeks, and 12 weeks
  Quality of life (QOL) will be evaluated by Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36).
Brain activation | Baseline, 8 weeks, and 12 weeks
  A multichannel wearable fNIRS imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NY, USA) will be used to detect the hemodynamics of brain areas associated with the agility test, cognitive tasks, and single and dual task walking test.

OTHER OUTCOMES:
Montreal Cognitive Assessment (MoCA) | Baseline, 8 weeks, and 12 weeks
  MoCA contains 16 items and 11 categories to assess multiple cognitive domains, is a screening instrument for MCI, and its validity has been established in various clinical groups and countries.
Working memory | Baseline, 8 weeks, and 12 weeks
  The backward digit span test (DGS) will be used to measure working memory.
Mental set shifting | Baseline, 8 weeks, and 12 weeks
  The Wisconsin Card Sorting Test (WCST) will be used to measure participants' ability to shift their cognitive ability in response to the demands of environment.
Selective attention and inhibition | Baseline, 8 weeks, and 12 weeks
  The Stroop Color and Word Test (SCWT) will be used to measure selective attention.
Motor Function | Baseline, 8 weeks, and 12 weeks
  Walking performance, normal walking, cognitive dual-task walking, muscle strength of bilateral lower limbs, five times sit to stand test, timed up and go, quiet static standing task, and the 360° turning task, flexibility, 6-minute walk test (6WMT)

CONTACTS AND LOCATIONS:
Overall Officials: Yan Ci Liu, PhD, Principal Investigator — National Taiwan University